CLINICAL TRIAL: NCT06663813
Title: Enhancing Proactive and Preventative Health Behaviors Among Hyperglycemic Patients Presenting to the Emergency Department
Brief Title: Enhancing Preventative Health Behaviors Among Emergency Department Hyperglycemic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Sara Heinert, PhD, MPH, Co-Director of Research; Assistant Professor at the Department of Emergency Medicine, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro2024000602
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Hyperglycemia
Keywords: Emergency Medicine; Type 2 Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants in the intervention arm will receive Type 2 Diabetes Mellitus educational materials that includes information regarding Type 2 Diabetes symptoms, risk factors, and resources for further follow-up care alongside standard Emergency Medicine care, which includes discharge instructions provided by ED practitioners along with verbal explanations from their assigned ED nurse.
  Interventions: Behavioral: Educational Intervention

INTERVENTIONS:
Behavioral: Educational Intervention — Utilizing the Health Belief model, educational materials detailing diabetes risk factors to address perceived susceptibility, diabetes severity and complications to address perceived severity, and PCP follow-up information and medication assistance programs to address perceived barriers will be provided.

SUMMARY:
The goal of this clinical trial is to increase Type 2 Diabetes Mellitus knowledge and awareness among patients who present to the Emergency Department with hyperglycemia. The main questions it aims to answer are:

* How do patients view their risk of developing type 2 diabetes based on their demographics and behaviors?
* Does giving patient education increase patient knowledge, leading to healthier behaviors?

Researchers will assess if the educational intervention increases diabetes knowledge and positive health behaviors among Emergency Department hyperglycemic patients.

Participants will:

* Receive the educational packet (intervention) alongside standard Emergency Care.
* Take pre-survey at time of Emergency Department visit and post- survey two weeks later.

DETAILED DESCRIPTION:
Despite the large prevalence of patients presenting to the Emergency Department (ED) with hyperglycemia or disease manifestations related to Type 2 Diabetes Mellitus (T2DM), there remains a gap in our understanding of rapid educational strategies delivered within the ED itself. As such, the goal of this project is to utilize the Health Belief Model (HBM) framework to target ED patients' perceived susceptibility, severity, benefits, and barriers in an effort to enhance proactive health behaviors, such as primary care physician (PCP) follow-up and utilization of medication assistance programs, among ED patients.

We will recruit 400 English speaking adults who present to the ED with a blood glucose of ≥200 mg/dL. All participants will receive educational materials on diabetes, as well as resources to local primary-care follow up and medication assistance programs. Participants will complete pre- and post-surveys to quantify changes in self-perceived susceptibility, severity, barriers to managing T2DM, and behavioral changes, which include presence of PCP follow-up, establishing a new PCP, and utilizing medication assistance programs.

Quantitative pre- and post-survey responses will be analyzed via regression models and paired t-tests to evaluate for statistically significant changes in perceived susceptibility, severity, benefits, and barriers to T2DM self-management among participants before and after receiving the educational intervention.The expected findings of this research study are increases in patient diabetes knowledge and self-perception of susceptibility and severity, leading to higher rates of PCP follow-up among participants following dissemination of educational materials grounded in the HBM framework. These research outcomes can be utilized to inform future interventions that target further barriers or reduce ED recidivism for hyperglycemic patients in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Persons 18 years of age or older who present as patients in the Robert Wood Johnson University Hospital Emergency Department with or without a preexisting Type 2 Diabetes Mellitus diagnosis with a blood glucose of ≥200 mg/dL. Participants must speak English to participate in the study.

Exclusion Criteria:

* Age less than 18 years and blood glucose <200 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Knowledge | Initial Emergency Department presentation to follow-up survey (2 weeks later)
  Changes in self-perceived susceptibility, severity, benefits, and barriers to managing T2DM, aligned with the Health Belief Model

SECONDARY OUTCOMES:
Proactive and Preventative Health Behaviors | Initial Emergency Department presentation to follow-up survey (2 weeks later)
  Behavioral changes, which include presence of PCP follow-up, establishing a new PCP, and utilizing medication assistance programs.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Heinert, PhD, MPH, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- One Robert Wood Johnson Place, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in this article, after deidentification (including text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Due to the nature of the data being collected, and to ensure participant confidentiality, data will be made available using a tiered request for access system. All tiers of data require a data-use agreement (DUA) at a minimum, additional precautions for restricted-use will be included in data request forms.

REFERENCES:
- See also: This research table demonstrates that T2DM is currently the most prevalent chronic disease encountered in the ED. — https://archive.cdc.gov/www_cdc_gov/nchs/data/ahcd/nhamcs_emergency/2010_ed_web_tables.pdf
- See also: Describes the tenants of the Health Belief Model — https://www.mheducation.co.uk/predicting-and-changing-health-behaviour-research-and-practice-with-social-cognition-models-9780335263783-emea-group